## **CONSENT (ENGLISH)**

## **Consent for Participation in the study**

I understand that a study "Effect of Patient Information Leaflet on working pattern and patient satisfaction level in a busy Indian day care operative theatre complex" conducted by Department of Anesthesia and Department of Head Neck surgery, involves filling of a questionnaire in the minor OT. The questionnaire includes questions with respect to the procedure planned/ done in minor OT. No personal details other than age, gender and educational details will be asked. Participation in this study is completely voluntary and it would take around 5 minutes to fill the feedback form

I understand that there would not be any additional medical procedures or any risk involved in participating in the trial. I understand that this study has been approved by the Institutional Ethics Committee, Tata Memorial Centre. The confidentiality with regard to my medical data will be ensured, and that the results published will not be linked to me. I understand that, if needed, the investigating team - **Dr S Bakshi, Dr A Panigrahi, Dr A Tambule, Dr P Pai**, contact no 022- 24177000 would be willing to provide any additional information regarding the study.

I understand that no payment will be made to me for participation and I am willing to allow the use of my data for the study.

I have read the above information. I have received a copy of this form.

| Participant's name : |
|---------------------------------|
| Participant's signature & date: |
| Address: |
| Name of PI or Co-PI/Co-I: |
| PI or Co-PI/Co-I & date: |

Version No. 1 05/11/2016